CLINICAL TRIAL: NCT03436953
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of CX-8998 for Tremor Associated With Parkinson's Disease
Brief Title: A Phase 2 Study of CX-8998 in Adults With Tremor Associated With Parkinson's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The program was not initiated nor were any patients ever enrolled. The investigations detailed in the submitted protocol were incorporated into another program.
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CX-8998-CLN2-003
Record Dates: First submitted 2018-02-07; First posted 2018-02-19 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Parkinson's Disease; Tremor
MeSH Terms: conditions — Parkinson Disease; Tremor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CX-8998 T-type calcium channel blocker (Experimental)
  Interventions: Drug: CX-8998
- Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CX-8998 — T-type calcium channel blocker
  Arms: CX-8998 T-type calcium channel blocker
Drug: Placebo — Placebo comparator
  Arms: Comparator

SUMMARY:
This is a Phase 2, multicenter, double-blind, placebo-controlled, parallel-group study consisting of a screening period of up to 4 weeks, a 4 week randomized double-blind, dose-titration treatment period, followed by a 1 week safety follow-up period after the last dose of study medication, and a scheduled follow-up safety telephone call one week later.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, double-blind, placebo-controlled, parallel-group study consisting of a screening period of up to 4 weeks, a 4 week randomized double-blind, dose-titration treatment period, followed by a 1 week safety follow-up period after the last dose of study medication, and a scheduled follow-up safety telephone call one week later.

Subjects will be randomized 1:1 to one of two treatment groups. Group A will receive titrating doses of CX-8998 up to 10 mg BID and Group B will receive placebo.

Subjects will participate for a total of up to 12 weeks, including screening, the 4-week treatment period and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Men or non-pregnant, non-breastfeeding women 40 to 80 years-of-age who are able to read and understand English.
* Mini Mental State Exam (MMSE) score ≥ 24.
* Clinical diagnosis of idiopathic Parkinson's disease and presence of at least 2 out of 3 cardinal characteristics (tremor, rigidity, and/or bradykinesia).
* Hoehn & Yahr Stage I III (inclusive) if not experiencing motor fluctuations. If experiencing motor fluctuations, must be Hoehn & Yahr Stage I IV (inclusive) when OFF or I-III (inclusive) when ON.
* An MDS-UPDRS tremor score (sum of items 2.10, 3.15, 3.16, 3.17, 3.18) of a least 10 (during ON for subjects experiencing fluctuations) (centrally rated) (Forjaz et al., 2015). A limited number of subjects with an MDS-UPDRS of 8 or 9 may be included with Sponsor approval.
* Treated with a stable regimen of anti-parkinsonian and/or anti-tremor medication (with the exception of primidone) for at least 2 weeks prior to screening. Changes to anti-parkinsonian or anti-tremor medications after screening is not permitted.

Exclusion Criteria:

* Current diagnosis of: a. essential tremor / b. cerebellar disease
* Presence or known history of: a. significant visual hallucinations (in the opinion of the Investigator and/or Study Safety Representative) / b. significant impulse control disorder (ICD) (in the opinion of the Investigator and/or Study Safety Representative).
* History or clinical features consistent with an atypical parkinsonian syndrome.
* Dyskinesia or dystonia that would, in the opinion of the investigator, central rater, or Sponsor, interfere with the assessment of tremor.
* Exposure to tremorigenic drugs or drug withdrawal states within the 30 days prior to the first planned dose of study drug.
* Direct or indirect trauma to the nervous system within 3 months preceding the onset of tremor.
* History or clinical evidence of psychogenic tremor origin. Known history of other medical or neurological conditions that may cause or explain subject's tremor.
* Prior MR-guided Focused Ultrasound or surgical intervention (e.g., deep brain stimulation, ablative thalamotomy or gamma knife thalamotomy) for treatment of tremor or Parkinson's disease.
* Use of medication(s) in the past month that might produce tremor or interfere with the evaluation of tremor.
* Inability to refrain from use of medication/substance(s) that might produce tremor or interfere with the evaluation of tremor on study visit days.
* Positive urine drug screen for drugs of abuse, except if this is explained by use of an allowed prescription medicine.
* Regular use of more than two units of alcohol per day.
* Use of prescription or non-prescription drugs or other products (i.e. grapefruit juice) known to be strong inhibitors or inducers of CYP3A4 which cannot be discontinued 2 weeks prior to Day 1 of dosing and withheld throughout the study.
* Concurrent illnesses that would be a contraindication to trial participation.
* Psychological, social, familial, or geographical reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.
* Any other condition and/or situation that causes the Investigator or Study Safety Representative to deem a subject unsuitable for the study (e.g., due to expected study medication non-compliance, inability to medically tolerate the study procedures, or a subject's unwillingness to comply with study-related procedures).
* Treatment with an investigational agent within 30 days prior to the first dose of CX-8998 or planning to receive an investigational agent during the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Day 28 on the MDS-UPDRS Tremor Score as scored by the central rater | Baseline through completion of study treatment period, an average of 28 days
  The MDS-UPDRS is a multi-dimensional scale that assesses the motor and non-motor impact of PD across four parts. Part I: Non-Motor Experiences of Daily Living; Part II: Motor Experiences of Daily Living; Part III: Motor Examination; and Part IV: Motor Complications.

SECONDARY OUTCOMES:
Change from Baseline to Day 28 on the TETRAS Activity of Daily Living subscale | Baseline through completion of study treatment period, an average of 28 days
  The ADL section of TETRAS has 12 items, each rated 0, 1, 2, 3 or 4. The maximum total score is 48. Item 1 addresses speech; item 10 addresses occupational impairment; and item 12 assesses social impact. The other 9 items assess activities that are affected primarily by upper limb tremor
Change from Baseline to Day 28 in accelerometry score | Baseline through completion of study treatment period, an average of 28 days
  Accelerometry will be used to obtain quantitative measurements of tremor. The Kinesia ONE device will be placed on the index finger and worn in the clinic immediately after execution of the MDS-UPDRS and/or TETRAS performance subscale. A total of 4 tasks will be performed on the left side and then again on the right side to assess resting, postural, kinetic, and lateral wing beating tremor. Each task will be performed for 15 seconds.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] as assessed by CTCAE v4.0 | Through study completion, an average of 12 weeks
  Treatment-emergent adverse events are all adverse events occurring during the treatment period or a pretreatment event that worsens in intensity during the treatment period.
Changes from baseline in QTcF | Baseline through study completion, an average of 5 weeks
  Fridericia's Correction Formula (QTCF) is a formula which takes into account the physiologic shortening of the QT interval which occurs as the heart rate increases, permitting comparison of the QT interval across a range of rates.
Percentage of subjects who did not complete the study due to Treatment Emergent Adverse Events as assessed by CTCAE v4.0 | Duration of study, an average of 12 weeks
  Treatment-emergent adverse events are all adverse events occurring during the treatment period or a pretreatment event that worsens in intensity during the treatment period.
Percentage of subjects with Serious Adverse Events as assessed by CTCAE v4.0 | Duration of study, an average of 12 weeks
  Any adverse event that results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect observed in any offspring of the subject conceived during treatment with the study drug or is an important medical event.
Percentage of subjects with Adverse Events of Special Interest as assessed by CTCAE v4.0 | Duration of study, an average of 12 weeks
  An adverse event of special interest is a serious adverse event as defined in Outcome 8.
Columbia-Suicide Severity Rating Scale (C-SSRS) | Screening through study completion, an average of 8 weeks
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a questionnaire used for suicide assessment. A numerical score is derived from the C-SSRS categories. The score is created at each assessment for each patient and is used for determining treatment emergence. Suicidal Ideation Score: The maximum suicidal ideation category (1-5 on the C-SSRS) present at the assessment.
Epworth Sleepiness Scale | Baseline through completion of study treatment period, an average of 28 days
  The Epworth Sleepiness Scale (ESS) is a scale intended to measure daytime sleepiness that is measured by use of a very short questionnaire. The questionnaire asks the subject to rate his or her probability of falling asleep on a scale of increasing probability from 0 to 3 for 8 different situations. The scores are added together to obtain a single number.
Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease-Rating Scale (QUIP-RS) | Screening through study completion, an average of 8 weeks
  The QUIP-RS was developed to assess the severity of impulse control disorders and related behavior symptoms and to monitor changes in symptoms over time. The QUIP-RS has 4 primary questions (pertaining to commonly reported thoughts, urges/desires, and behaviors associated with impulsive control disorders), each of which is applied to 4 impulsive behaviors (compulsive gambling, buying, eating, and sexual behavior) and 3 related disorders (medication use, punding, and hobbyism). It uses a 5-point scale to gauge the frequency of behaviors. Scores for each behavior and related disorder range from 0 to 16, with a higher score indicating greater severity (ie, frequency) of symptoms. The total QUIP-RS score for all impulsive control disorders and related disorders combined ranges from 0 to 112.
University of Miami Parkinson's disease Hallucinations Questionnaire (UM-PDHQ) | Screening, Baseline and Day 28, an average of 28 days
  The UM-PDHQ is a 20-item clinician-administered questionnaire that is completed during a structured interview. Questions are divided into 2 groups: a quantitative group that consists of 6 questions (modality, frequency, duration, insight, emotional burden) and a qualitative group that consists of 14 questions. Scores range from 0-14.
Hospital Anxiety and Depression Scale (HADS) | Screening and Day 28, an average of 28 days
  The Hospital Anxiety and Depression Scale (HADS), a self-assessment scale, was developed to detect states of depression, anxiety and emotional distress. The HADS is a 14-item scale that generates ordinal data. Seven of the items relate to anxiety, and 7 of the items relate to depression. Each item on the questionnaire is scored from 0 to 3, with individual scores ranging between 0 and 21 for either anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Boyer, PhD, Study Director — Jazz Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Undecided